CLINICAL TRIAL: NCT05287126
Title: An Open-Label, Single-Arm Study to Evaluate the Efficacy, Pharmacokinetics, and Safety of Etrasimod in Adolescent Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate Etrasimod Treatment in Adolescents With Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD334-207; C5041010 (Other: Alias Study Number); 2022-500345-25-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06025227 (Available)
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
Keywords: Pharmacokinetics; Adolescents; Active Ulcerative Colitis; APD334
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etrasimod (Experimental)
  Interventions: Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — Etrasimod tablet or granules by mouth, once daily up to 52 weeks of treatment.
  Other Names: APD334

SUMMARY:
The purpose of this study is to determine the safety, efficacy, and pharmacokinetics (PK) of etrasimod for the treatment of moderately to severely active ulcerative colitis in adolescents (≥ 12 years up to < 18 years of age). Participants who will complete the total 52-week treatment period will have the opportunity to continue in a Long-Term Extension (LTE) Period of up to 4 years (5 years after study enrollment).

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of ulcerative colitis (UC) that is moderately to severely active
* Participants are permitted to be receiving a therapeutic dose of select UC therapies

Exclusion criteria:

* Severe extensive colitis
* Diagnosis of Crohn's disease (CD) or indeterminate colitis or the presence or history of a fistula consistent with CD
* Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2027-07-14 (Estimated); Study Completion 2031-08-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Clinical Remission as Assessed by Modified Mayo Score (MMS) at Week 52 | Week 52

SECONDARY OUTCOMES:
Plasma Concentration of Etrasimod at 4 Hours Post-dose (C4h) | 4 hours (± 15 minutes) post-dose
Plasma Steady State Trough Concentration (Ctrough,ss) of Etrasimod | pre-dose and 4 hours (±15 minutes) post-dose at Day 1; at trough concentrations (approximately 24 hours after the dose taken the day before the study visit) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Proportion of Participants Achieving Clinical Remission as Assessed by MMS at Week 12 | Week 12
Proportion of Participants Achieving Endoscopic Improvement at Week 12 | Week 12
Proportion of Participants Achieving Endoscopic Improvement at Week 52 | Week 52
Proportion of Participants Achieving Symptomatic Remission at Week 12 | Week 12
Proportion of Participants Achieving Symptomatic Remission at Week 52 | Week 52
Proportion of Participants with Clinical Remission at Week 12 Who Had Not been Receiving Corticosteroids for ≥ 2 weeks Prior to Week 12 | Week 12
Proportion of Participants with Clinical Remission at Week 52 Who Had Not been Receiving Corticosteroids for ≥ 12 weeks Prior to Week 52 | Week 52
Proportion of Participants Achieving Clinical Response at Week 12 | Week 12
Proportion of Participants Achieving Clinical Response at Week 52 | Week 52
Proportion of Participants Achieving Clinical Remission by Pediatric Ulcerative Colitis Activity Index (PUCAI) at Week 12 | Week 12
Proportion of Participants Achieving Clinical Remission as Assessed by PUCAI at Week 52 | Week 52
Proportion of Participants Achieving a Clinical Response as Assessed by PUCAI at Week 12 | Week 12
Proportion of Participants Achieving a Clinical Response as Assessed by PUCAI at Week 52 | Week 52
Number and Severity of Adverse Events | Up to Week 52
  Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- United States (20):
  - Arkansas Children's (IP Address), Little Rock, Arkansas
  - Arkansas Children's, Little Rock, Arkansas
  - Valley View Wellness Medical Center, Garden Grove, California
  - Loma Linda Children's Hospital, Loma Linda, California
  - Loma Linda University Clinical Trial Center, Loma Linda, California
  - Loma Linda University Eye Institute, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda University Pediatric Clinics, Loma Linda, California
  - Loma Linda University Children's Hospital Pediatric Specialty Clinics, San Bernardino, California
  - University of California San Francisco,, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - University of California,San Francisco Pediatric ClinicalResearch Center (PCRC), San Francisco, California
  - Arnold Palmer Hospital - Center for Digestive Health and Nutrition, Orlando, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - William Beaumont Hospitals Reference Laboratory, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University Hospitals Cleveland Medical Center Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Advance Clinical Trial PLLC, Abilene, Texas
- Landeskrankenhaus Salzburg, Salzburg, Austria
- University Hospitals Leuven, Leuven, Belgium
- Japan (11):
  - Tsujinaka Hospital - Kashiwanoha, Kashiwa, Chiba
  - Ishii Eye Clinic, Nagareyama-shi, Chiba
  - Gunma University Hospital, Maebashi, Gunma
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kinki University - Nara Hospital, Ikoma, Nara
  - Saitama Prefectural Children's Medical Center, Saitama-shi, Saitama
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Saga University Hospital, Saga
  - Toyama Prefectural Central Hospital, Toyama
- Poland (8):
  - WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Masovian Voivodeship
  - Instytut "Pomnik - Centrum Zdrowia Dziecka" (IPCZD) (The Children's Memorial Health Institute), Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - Twoja Przychodnia - Szczecińskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Slovakia (2):
  - Narodny ustav detskych chorob, Bratislava, Bratislava Region
  - Cliniq s.r.o., Bratislava
- Spain (4):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Consorci Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-207